CLINICAL TRIAL: NCT03394209
Title: An Adaptive Study of the Pharmacokinetics of Favipiravir in Patients With Severe
Brief Title: A Pharmacokinetics Study of Favipiravir in Patients With Severe Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Institute of Pharmacology and Toxicology (Other); University of Oxford (Other); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Bin Cao, Dr.Bin Cao, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAVI-PK-2017001
Record Dates: First submitted 2017-12-25; First posted 2018-01-09 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Influenza, Human; Critical Illness; Influenza
Keywords: Favipiravir, Influenza, Human, Critical Illness, Pharmacokinetics
MeSH Terms: conditions — Influenza, Human; Critical Illness | interventions — favipiravir; Oseltamivir

STUDY DESIGN:
Intervention Model Description: This is a adaptive study, which include two steps.
  1st step: 1600mg BID on day 1, followed by 600mg BID for 9 days. Sample size: 15 PK analysis: If the proportion of patients with a minimum observed plasma trough concentration above the MEC (20μg/ml) at all measured time points after the second dose is greater than or equal to 80% then the dose is considered adequate and the study will be completed. If not, then a second patient cohort will be recruited and will receive favipiravir 1800mg BID on day 1, followed by favipiravir 800mg BID for 9 days. Sample size: 15
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Favipiravir+oseltamivir (Experimental): Favipiravir+oseltamivir will be given twice daily for a 10-day period.
  Interventions: Drug: Favipiravir; Drug: Oseltamivir 75Mg Capsule

INTERVENTIONS:
Drug: Favipiravir — In first step: favipiravir tablet is orally administered. This drug will be given twice daily for a 10-day period. For the First day, the dosage is 1600 mg twice daily. Starting from the second day, the dosage is 600 mg twice daily.
  In second step: favipiravir tablet is orally administered. This drug will be given twice daily for a 10-day period. For the First day, the dosage is 1800 mg twice daily. Starting from the second day, the dosage is 800 mg twice daily.
  Other Names: T-705
Drug: Oseltamivir 75Mg Capsule — oseltamivir will be administered at 75mg twice daily orally for 10 days

SUMMARY:
Title: An adaptive study of the pharmacokinetics of favipiravir in patients with severe influenza Study Design: An open label, single group assignment, adaptive study to evaluate the pharmacokinetics of favipiravir in adult patients with severe influenza.

In the first stage, participants will receive favipiravir 1600mg BID on day 1, followed by favipiravir 600mg BID for 9 days.

If the proportion of patients with a minimum observed plasma trough concentration above the MEC (20μg/ml) at all measured time points after the second dose is less than 80% then a second patient cohort will be recruited and will receive favipiravir 1800mg BID on day 1, followed by favipiravir 800mg BID for 9 days.

Intervention: The 1st stage: 1600mg BID on day 1, followed with 600mg BID for 9 days. Sample size: 15 The 2nd stage: 1800mg BID on day 1, followed with 800mg BID for 9 days. Sample size: 15 Population: Males and females aged 18 years or older admitted to hospital with a positive PCR test for influenza and a PaO2/FiO2≤300mmHg or/and on mechanical ventilation for severe lung infection on admission.

Sample size 15 or 30 severe influenza patients Research hypothesis The administration of oral favipiravir at either 1600mg/600mg BID or 1800/800mg BID will result in ≥ 80% patients achieving a minimum observed plasma trough concentration above the MEC (20μg/ml) at all measured time points after the second dose.

Phase: Phase 2a, PK, safety and feasibility study. Description of Study Agent: Favipiravir (T-705) a viral RNA-dependent RNA polymerase inhibitor.

Study Duration: 1 year Participant Duration: 38 days

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized males or females with a positive PCR test for influenza virus infection
2. Adults aged ≥18years
3. PaO2/FiO2≤300mmHg or on mechanical ventilation
4. < 10 days since symptom onset
5. Negative pregnancy testing for childbearing age females (under 60 years)
6. Willingness to use contraception for 7 days after end of treatment
7. Informed consent
8. In addition, male subjects must:

   1. Agree not to donate sperm during the study and for 7 days following the last dose of study drug, and
   2. Agree to adhere strictly to one of the following contraceptive measures from the Screening Visit until 7 days after the last dose of study drug:

   i. abstain from sexual intercourse or ii. have a female partner using effective means of birth control as noted below or iii. use a condom with spermicide or a second barrier method by female partner.

Female subjects

a. Of child-bearing potential must agree to adhere strictly to one of the following approved contraceptive measures during the study and for 7 days after the last dose of study drug: i. abstain from sexual intercourse or ii. have a male partner incapable of fathering a child (eg, had a vasectomy at least 6 months with history of negative semen analysis prior Screening or iii. use of one of the following methods, in combination with condom and spermicide use by a male partner: nonhormonal intrauterine device (IUD); diaphragm; or hormonal contraceptives including oral contraceptives, injectable subdermal implants, hormonal IUD, or vaginal ring b. Be unable to bear children defined as one of the following: i. absence of a menstrual period for ≥12 consecutive months with FSH confirmation, ii. be 60 years of age or greater, iii. had surgical removal of uterus or removal of both ovaries, or iv. had undergone tubal ligation >6 weeks prior to Day 1 dosing

Exclusion Criteria:

1. Any condition that does not allow for safely following the protocol
2. Patient refusal to accept invasive organ support treatment if needed
3. Pregnant or breastfeeding
4. Any condition resulted to reception of renal replacement therapy
5. AST > 5 times upper of limit or Child Pugh score ≥ C
6. Serum uric acid level > 3 times upper level of normal (430 ummol/L) associated with symptoms of gout
7. Has a history of gout or is under treatment for: gout or hyperuricemia; hereditary xanthinuria; hypouricemia or xanthine calculi of the urinary tract
8. Has a history of hypersensitivity to an anti-viral nucleoside-analog drug targeting a viral RNA polymerase
9. Physician makes a decision that trial involvement is not in patients' best interest.
10. Currently or have been involved in another anti-influenza treatment trial in the last 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with minimum plasma of Favipiravir trough concentration above the MEC (20μg/ml) at all measured time points after the second dose. | 10 days during the intervention period

SECONDARY OUTCOMES:
Maximum plasma concentration observed over the treatment period (Cmax ) | 10 days during the intervention period
Minimum plasma concentration observed over the treatment period (Cmin) | 10 days during the intervention period
Average pre-dose plasma concentration (Trough) | 10 days during the intervention period
Proportion of patients whose favipiravir plasma concentration at least one time exceeds MEC in study days | 10 days during the intervention period
The proportion of patients falling into each category of a five-point ordinal scale on day 10 and day 28 after starting favipiravir | 28 days from starting intervention
  The category of a five-point ordinal scale: death; hospitalised on ECMO and/or mechanical ventilation; hospitalised on supplemental oxygenation; hospitalised not on supplemental oxygenation; discharged.
Duration (days) of mechanical ventilation | from reception of mechanical ventilation to ventilator weening, an average of 10 days
Duration (days) of extracorporeal membrane oxygenation | from starting ECMO to weening, an average of 9 days
Duration (days) of supplemental oxygenation | Duration (days) of hospitalization with oxygen therapy，an average of 13 days
Duration (days) of hospitalization | Days from admission to discharge，an average of 19 days
The proportion of patients with a negative RT-PCR for influenza from upper and/or lower respiratory tract samples on day 10 after starting treatment | Duration of viral shedding,an average of 15 days
The time (days) to negative RT-PCR for influenza from upper and/or lower respiratory tract samples (capped at day 10) | Duration of viral shedding,an average of 15 days
The proportion of patients with drug related adverse events | 38 days from starting intervention
The proportion of patients with genetic and phenotypic markers of resistance to favipiravir and/or oseltamivir | Days from admission to discharge，an average of 19 days

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gao HN, Lu HZ, Cao B, Du B, Shang H, Gan JH, Lu SH, Yang YD, Fang Q, Shen YZ, Xi XM, Gu Q, Zhou XM, Qu HP, Yan Z, Li FM, Zhao W, Gao ZC, Wang GF, Ruan LX, Wang WH, Ye J, Cao HF, Li XW, Zhang WH, Fang XC, He J, Liang WF, Xie J, Zeng M, Wu XZ, Li J, Xia Q, Jin ZC, Chen Q, Tang C, Zhang ZY, Hou BM, Feng ZX, Sheng JF, Zhong NS, Li LJ. Clinical findings in 111 cases of influenza A (H7N9) virus infection. N Engl J Med. 2013 Jun 13;368(24):2277-85. doi: 10.1056/NEJMoa1305584. Epub 2013 May 22. PMID 23697469
- [Result] Zheng S, Tang L, Gao H, Wang Y, Yu F, Cui D, Xie G, Yang X, Zhang W, Ye X, Zhang Z, Wang X, Yu L, Zhang Y, Yang S, Liang W, Chen Y, Li L. Benefit of Early Initiation of Neuraminidase Inhibitor Treatment to Hospitalized Patients With Avian Influenza A(H7N9) Virus. Clin Infect Dis. 2018 Mar 19;66(7):1054-1060. doi: 10.1093/cid/cix930. PMID 29077848
- [Result] Li H, Yang SG, Gu L, Zhang Y, Yan XX, Liang ZA, Zhang W, Jia HY, Chen W, Liu M, Yu KJ, Xue CX, Hu K, Zou Q, Li LJ, Cao B, Wang C; National Influenza A(H1N1)pdm09 Clinical Investigation Group of China. Effect of low-to-moderate-dose corticosteroids on mortality of hospitalized adolescents and adults with influenza A(H1N1)pdm09 viral pneumonia. Influenza Other Respir Viruses. 2017 Jul;11(4):345-354. doi: 10.1111/irv.12456. Epub 2017 Jun 9. PMID 28464462
- [Result] Wang X, Jiang H, Wu P, Uyeki TM, Feng L, Lai S, Wang L, Huo X, Xu K, Chen E, Wang X, He J, Kang M, Zhang R, Zhang J, Wu J, Hu S, Zhang H, Liu X, Fu W, Ou J, Wu S, Qin Y, Zhang Z, Shi Y, Zhang J, Artois J, Fang VJ, Zhu H, Guan Y, Gilbert M, Horby PW, Leung GM, Gao GF, Cowling BJ, Yu H. Epidemiology of avian influenza A H7N9 virus in human beings across five epidemics in mainland China, 2013-17: an epidemiological study of laboratory-confirmed case series. Lancet Infect Dis. 2017 Aug;17(8):822-832. doi: 10.1016/S1473-3099(17)30323-7. Epub 2017 Jun 2. PMID 28583578
- [Result] Dunning J, Baillie JK, Cao B, Hayden FG; International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC). Antiviral combinations for severe influenza. Lancet Infect Dis. 2014 Dec;14(12):1259-70. doi: 10.1016/S1473-3099(14)70821-7. Epub 2014 Sep 8. PMID 25213733
- [Result] Kumar A. Early versus late oseltamivir treatment in severely ill patients with 2009 pandemic influenza A (H1N1): speed is life. J Antimicrob Chemother. 2011 May;66(5):959-63. doi: 10.1093/jac/dkr090. Epub 2011 Mar 15. PMID 21406435
- [Result] Kile JC, Ren R, Liu L, Greene CM, Roguski K, Iuliano AD, Jang Y, Jones J, Thor S, Song Y, Zhou S, Trock SC, Dugan V, Wentworth DE, Levine MZ, Uyeki TM, Katz JM, Jernigan DB, Olsen SJ, Fry AM, Azziz-Baumgartner E, Davis CT. Update: Increase in Human Infections with Novel Asian Lineage Avian Influenza A(H7N9) Viruses During the Fifth Epidemic - China, October 1, 2016-August 7, 2017. MMWR Morb Mortal Wkly Rep. 2017 Sep 8;66(35):928-932. doi: 10.15585/mmwr.mm6635a2. PMID 28880856